



An Evaluation of an ACT and PBS Group for Parents and Education Staff of Children and Young People with an Intellectual Disability Education Staff Consent Form (non-CTIMP/CE device), version no. 2, 17/12/2018

## **Consent Form (version 2)**

## An Evaluation of an ACT and PBS Group for Parents and Education Staff of Children and Young People with an Intellectual Disability

| Participant ID: | | | | |
|---|---|---|---|---|
| | | | Initial here for YES | Initial here for NO |
| 1. I confirm that I have read and understa | nd the information sheet | | | |
| (Education Staff PIS version 2, 17.12.2018) for the above study and have | | | | |
| had the opportunity to consider the information for a minimum of 24 hours | | | | |
| and ask questions. | | | | |
| 2. I understand that my participation is vol | untary and that I am free to | | | |
| withdraw at any time, without giving any reason, without my medical care or | | | | |
| legal rights being affected. | | | | |
| 3. I understand that relevant sections of da | ata collected during the stud | dy may | | |
| be looked at by individuals from the regulatory authorities and from the | | | | |
| Sponsors (NHS Lothian and the University of Edinburgh) or from the/other | | | | |
| NHS Board(s) where it is relevant to my ta | aking part in this research. I | give | | |
| permission for those individuals to have access to my records. | | | | |
| 4. I agree to my General Practitioner (GP) being informed of my participation | | | | |
| in this study. | | | | |
| 5. I agree to a summary of the study results being sent to me by post. | | | | |
| 6. I agree to the focus group being audio-recorded, for the purposes of | | | | |
| allowing it to be transcribed. | | | | |
| 7. I agree to take part in the above study. | | | | |
| Name of Participant | Date | Signatu | re | |
| Name of Person taking consent | Date | <br>Signatu | re | |

1x original – into Site File; 1x copy – to Participant;